CLINICAL TRIAL: NCT06387927
Title: The Effectiveness of Home-based Exercise Programs Versus Supervised Conventional Core Stability Exercises in Treatment of Chronic Mechanical, Non-specific Low Back Pain Patients With Controlled Hypertension
Brief Title: Effect of Home-exercise Programs Versus Supervised Core Stability Exercises on Hypertensive Patient With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Ababa, lecturer, Ahram Canadian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PT-NEUR-10/2023-520
Record Dates: First submitted 2024-04-19; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Hypertension; Low Back Pain
MeSH Terms: conditions — Hypertension; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (control) received supervised conventional core stability exercise program Study (Active Comparator): Group A (control) received supervised conventional core stability exercise program
  Interventions: Other: the core stability exercise
- group B received a home-based exercise program (Experimental): Group B received a home-based exercise program.
  Interventions: Other: home exercise program

INTERVENTIONS:
Other: home exercise program — Patients in group B were taught the core stability exercise in the first visit they received Arabic printed booklet for exercise description repetitions with diagrams in addition to Arabic illustration videos, they received a weekly telephone call to ensure their compliance to the exercise & motivation.
  Arms: group B received a home-based exercise program
Other: the core stability exercise — supervised conventional core stability exercise
  Arms: Group A (control) received supervised conventional core stability exercise program Study

SUMMARY:
Thirty male and female hypertension patients with chronic mechanical non-specific low back pain were included in this randomized controlled study conducted at the Ababa Private Physical Therapy Center in Beni-Seuf, Egypt. They were randomly assigned into two equal groups; the study group A control (n = 15) had a supervised conventional core stability, while the study group B (n = 15) received a home exercise program. In both groups' patients had evaluations before and after their six-week course of therapy. Modified-modified Schober test was used to assess the active back range of motion (ROM), Arabic version of Oswestry disability index (ODI) was utilized to evaluate functional disability, and visual analog scale (VAS) was used to measure pain.

ELIGIBILITY:
Inclusion Criteria:

* hypertensive patient
* patient with chronic back pain
* The patients aged 30 to 50 years

Exclusion Criteria:

* Patients with vertebral fractures
* patient with surgical spinal fixation
* patient with rheumatic disorders
* patient with systemic diseases
* patient with multiple sclerosis.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-02 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Assessment of pain | up to 4 weeks
  Pain was assessed using the visual analog scale
Assessment of lumbar flexion range of motion | up to 4 weeks
  performed by modified modified schober test
Assessment of functional disability | up to 4 weeks
  performed by Oswestry disability questionnaire version 2.0

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No